CLINICAL TRIAL: NCT05298007
Title: Intervention Effect of High Definition Transcranial Direct Current Stimulation (HD-tDCS) on Anxiety Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Director of medical psychological department, Anhui Medical University, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ahmu-tdcs-anxiety
Record Dates: First submitted 2022-02-13; First posted 2022-03-28 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Transcranial Direct Current Stimulation; Anxiety; Magnetic Resonance Imaging
Keywords: Transcranial Direct Current Stimulation; Anxiety; Magnetic Resonance Imaging
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real stimulation (Active Comparator): Participants will receive active tDCS once daily for two weeks. The anode was placed over Fz with return electrodes placed at Fpz, Cz, F3 and F4. Fourteen2-mA sessions (ramp-up and ramp-down periods of 30 and 30 seconds, respectively) were applied for 20 minutes each day over 14 consecutive sessions.
  Interventions: Device: High definition transcranial direct current stimulation
- sham stimulation (Sham Comparator): Participants will receive sham tDCS once daily for two weeks. Sham HD-tDCS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.
  Interventions: Device: sham high definition transcranial direct current stimulation

INTERVENTIONS:
Device: High definition transcranial direct current stimulation — tDCS is described as a non-invasive form of brain stimulation that uses a low-intensity, constant current applied directly to the head through scalp electrodes.
  Arms: real stimulation
Device: sham high definition transcranial direct current stimulation — Sham HD-tDCS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.
  Arms: sham stimulation

SUMMARY:
To investigate the intervention effect of high definition transcranial direct current stimulation (HD-tDCS) on anxiety symptoms and somatic symptoms in patients with anxiety disorder and its underlying neural mechanism by MRI.

DETAILED DESCRIPTION:
Anxiety is characterized by excessive fear, anxiety, or avoidance of a range of external and internal stimuli. Somatic symptoms often co-occur with anxiety and are part of the manifestation of anxiety. The purpose of this study was to explore the relieving effect of high definition transcranial direct current stimulation (HD-tDCS) on the symptoms of anxiety.

60 patients with anxiety disorder diagnosed by DSM-5 were recruited from the fourth people's Hospital of Hefei and the first affiliated Hospital of Anhui Medical University. All participants underwent a structured interview and routine laboratory examination before and after receiving HD-tDCS. After meeting the inclusion criteria and obtaining informed consent, each participant will complete the clinical evaluation, functional magnetic resonance imaging (fMRI) and HD-tDCS treatment conducted by trained researchers at the Neuropsychological Synergetic Innovation Center of Anhui Medical University. All the participants were randomized (1:1) to receive "active" or "sham" treatment protocol. The anode was placed over Fz with return electrodes placed at Fpz, Cz, F3 and F4. Fourteen 2-mA sessions (ramp-up and ramp-down periods of 30 and 30 seconds, respectively) were applied for 20 minutes each day over 14 consecutive sessions. Sham HD-tDCS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.

Before and after the HD-tDCS treatment, the patients had receiving a battery measure of neuropsychological tests and Magnetic resonance imaging scan in multimodalities. Neuropsychological assessment included MoCA, Stroop Test, VFT, DST, AVLT, HAMD, HAMA, PHQ15, BSS(Beck scale for suicide ideation),ISI,SDS, RRS, TEPS, AES, FPQ, PVAQ and AAS. Multimodal fMRI includes 3D-T1, rs-fMRI, DTI and ASL.

Neuropsychological evaluation and magnetic resonance imaging data were obtained again 24 hours after the last treatment. The symptoms of the patients were followed up one month after the end of treatment.They were instructed to focus their answers on the past week. Afterwards, they were unblinded by the study coordinator.

ELIGIBILITY:
Inclusion Criteria:

* the patients were diagnosed by more than 2 psychiatrists and met the diagnostic criteria of DSM-5 for anxiety, and HAMA>14, PHQ-15>5.
* the age ranged from 18 to 60 years old, and the length of education was more than 5 years.
* the visual acuity or corrected visual acuity is normal, right-handed, can cooperate with the completion of various experimental tests.

Exclusion Criteria:

* accompanied by severe somatic diseases, such as severe heart, liver, renal insufficiency and so on.
* accompanied by other neurological diseases, such as stroke, epilepsy and so on.
* pregnant and lactating women.
* accompanied by other mental disorders, such as drug abuse, schizophrenia, schizophrenic affective disorder, hysteria, autism and so on.
* patients with MRI taboos or factors affecting imaging quality, such as cardiac pacemaker, cochlear implant, cardio-cerebrovascular metal stent, metal denture, etc.
* those who could not cooperate with those who completed the relevant experiments, such as patients with depressive stupor, claustrophobia and so on.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
anxiety symptoms | baseline and immediately after intervention
  the change of anxiety symptoms assessed by HAMA scale(Hamilton Anxiety Scale) will constitute the major research outcome measure, to assess response to dDCS. HAMA scale scores range from 0 to 56 points, the higher the score indicates the more serious anxiety symptoms
resting-state functional connectivity | baseline and immediately after intervention
  the change of resting-state functional connectivity strength between stimulated target and the whole brain areas will be measured by functional MRI.

SECONDARY OUTCOMES:
somatic symptoms | baseline and immediately after intervention
  the change of somatic symptoms will be assessed by Patient Health Questionnaire (PHQ-15). PHQ-15 is composed of 15 physical symptoms that have been extracted from the PHQ. PHQ-15 scale scores range from 0 to 30 points. Higher scores indicate more severe somatic symptoms.
ISI(The insomnia severity index) | baseline and immediately after intervention
  ISI(The insomnia severity index) is used to evaluate the changes of sleep status of anxiety patients in the recent (2 weeks), which is a self-rating scale. ISI scale scores range from 0 to 28 points. The higher the score is, the worse the sleep quality is. This scale indirectly reflects the changes of patients' anxiety state through evaluation.
SAS(Self-rating anxiety scale) | baseline and immediately after intervention
  Self-rating anxiety scale(SAS) is a supplementary evaluation of the change of anxiety state of patients in this experiment, and it also belongs to the category of self-rating scale. Patients assessed anxiety by checking the frequency of 20 items: none or almost none, sometimes, most of the time, most of the time, or all of the time. SAS scale scores range from 0 to 100 points。The higher the score, the more serious the anxiety symptoms.
4DSQ-Som(Four-DimensionalSymptomQuestionnaire) | baseline and immediately after intervention
  The Four-DimensionalSymptomQuestionnaire (4DSQ) includes self-rating scale for depression, anxiety and somatization. In this experiment, only part of the somatization scale was used to evaluate the change of severity of patients' somatization symptoms. Patients need to check the frequency of 15 symptoms, the higher the score, the more severe the symptoms. 4DSQ-Som scale scores range from 0 to 60 points
HAMD(Hamilton Depression Scale) | baseline and immediately after intervention
  Anxiety patients are often complicated with depressive symptoms.The changes of depressive symptoms will assessed by HAMD, constituting the secondary research outcome. Hamilton Depression Scale (HAMD) compiled by Hamilton in 1960, is the most common clinical to assess Depression Scale. In this study, 17 versions were selected, and there were 17 questions. The subjects were assessed for their depression in the past week. Each question scored between 0 and 4 points.HAMD scale scores range from 0 to 54 points. Higher scores indicate more depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Zhang, Study Chair — Anhui Medical University
Locations (1):
- Anhui Medical University, Hefei, China